CLINICAL TRIAL: NCT05985590
Title: A Phase 1, Open-label, Fixed-sequence Study to Investigate the Effects of Multiple Doses of BMS-986278 on the Pharmacokinetics of Combined Oral Contraceptives (Drospirenone/Ethinyl Estradiol) in Healthy Female Participants
Brief Title: A Study to Investigate the Effects of BMS-986278 on Drospirenone and Ethinyl Estradiol Drug Levels in Healthy Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM027-1013
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; BMS-986278; Hormonal contraceptives; Ethinyl estradiol; Drospirenone; Pulmonary fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: DRSP/EE (Experimental)
  Interventions: Drug: Drospirenone/Ethinyl Estradiol
- Treatment B: BMS-986278/DRSP/EE (Experimental)
  Interventions: Drug: BMS-986278; Drug: Drospirenone/Ethinyl Estradiol

INTERVENTIONS:
Drug: BMS-986278 — Specified dose on specified days
  Arms: Treatment B: BMS-986278/DRSP/EE
Drug: Drospirenone/Ethinyl Estradiol — Specified dose on specified days

SUMMARY:
The purpose of the study is to assess the effects of BMS-986278 on Drospirenone (DRSP) and Ethinyl Estradiol (EE) when administered as a combined oral contraceptive in healthy female participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.0 and 32.0 kilograms/meter square (kg/m^2), inclusive.
* Body weight ≥ 45 kg.
* Healthy females, as determined by physical examination and clinical laboratory assessments (including chemistry, hematology, coagulation, and urinalysis) within the normal range at the screening visit and on Day -1, as applicable.

Exclusion Criteria:

* Any significant acute or chronic medical illness.
* Any gastrointestinal (GI) disease or surgery (including cholecystectomy) or other procedures (eg, bariatric procedures) that could affect drug absorption, distribution, metabolism, and excretion. Note: Appendectomy is allowed (12 months prior to screening).
* Any other clinically significant medical, psychiatric, and/or social reason, or other active issues, especially eye issues, as determined by the investigator.

Note: Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Predose and post-dose up to Day 28
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC [0-T]) | Predose and post-dose up to Day 28
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC [INF]) | Predose and post-dose up to Day 28

SECONDARY OUTCOMES:
Time of maximum observed concentration (Tmax) | Predose and post-dose up to Day 28
Terminal half-life (T-Half) | Predose and post-dose up to Day 28
Apparent total body clearance after extravascular administration (CL/F) | Predose and post-dose up to Day 28
Number of Participants with Adverse Events (AEs) | Up to Day 53
Number of Participants with Serious AEs (SAEs) | Up to Day 53
Number of Participants with AEs leading to discontinuation | Up to Day 53
Number of Participants with Physical Examination Abnormalities | Up to Day 28
Number of Participants with Vital Sign Abnormalities | Up to Day 28
Number of Participants with Electrocardiogram (ECG) Abnormalities | Up to Day 28
Number of Participants with Clinical Laboratory Abnormalities | Up to Day 27

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0002, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com